CLINICAL TRIAL: NCT05472805
Title: The Relationship of Neutrophil-Lymphocyte Ratio and Platelet-Lymphocyte Ratio to Carotid Intima-Media Thickness in Chronic Kidney Disease Patients Undergoing Dialysis
Brief Title: Neutrophil-Lymphocyte Ratio and Platelet-Lymphocyte Ratio to Predict Carotid Intima-Media Thickness in Chronic Kidney Disease Patients
Status: Completed | Type: Observational
Sponsor: Universitas Sebelas Maret (Other)
Responsible Party: Principal Investigator, Nurhasan Agung Prabowo, MD, Universitas Sebelas Maret
Other Study IDs: NLRandPLRtoCIMTinCKD
Record Dates: First submitted 2022-07-21; First posted 2022-07-25 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: Chronic Kidney Diseases; Dialysis; Complications; Coronary Heart Disease
Keywords: neutrophil-lymphocyte ratio; platelet-lymphocyte ratio; carotid intima-media thickness; chronic kidney disease; dialysis
MeSH Terms: conditions — Renal Insufficiency, Chronic; Coronary Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CIMT ≥1mm: The measurement of CIMT will be carried by a cardiologist in the cardiovascular department using B mode ultrasound. The cardiologist will measure both of the carotid artery, and higher measurement of CIMT will be recorded. This group includes individual with CIMT ≥1mm
- CIMT <1mm: The measurement of CIMT will be carried by a cardiologist in the cardiovascular department using B mode ultrasound. The cardiologist will measure both of the carotid artery, and higher measurement of CIMT will be recorded. This group includes individual with CIMT <1mm

SUMMARY:
This study aims to determine whether the neutrophil-lymphocyte ratio (NLR) and platelet-lymphocyte ratio (PLR) can be used as predictors of coronary heart disease (CHD) in CKD patients undergoing dialysis at Moewardi General Hospital Surakarta. It was hypothesized that NLR and PLR, which have been identified as inflammatory biomarkers, would be significantly related to increased arotid intima-media thickness (CIMT) in CKD patients undergoing dialysis. This study is an observational analytic study using a cross-sectional approach conducted at department of renal-hypertension and hemodialysis unit in Moewardi General Hospital in Surakarta, Indonesia from January to July 2022.

DETAILED DESCRIPTION:
This study is an observational analytic study using a cross-sectional approach conducted at department of renal-hypertension and hemodialysis unit in Moewardi General Hospital in Surakarta, Indonesia from January to July 2022. All patients aged 18 years old or older, with a diagnosis of CKD stage V and on HD or CAPD based RRTs were included in the study. The presence of cardiovascular, neoplastic, chronic inflammatory, or infectious disease, and usage of immunosuppressants or antiplatelet drugs precludes the patient from participating in the study.

The main outcome in this study is the presence of a high risk of CHD characterized by CIMT ≥1 mm. The risk of CHD will be operated as categorical variable; CIMT <1 mm and CIMT ≥1 mm. The main predictors used in this study are NLR and PLR. The absolute values of neutrophils and platelets were divided by the absolute values of lymphocytes to get the NLR and PLR values, respectively. Several confounding variables were also considered, including age, gender, nutrition status, CKD duration, presence of diabetes mellitus, and other hematologic parameters. These hematologic parameters include hemoglobin, leukocyte count, platelet count, neutrophils, and lymphocytes. These predictors will be operated as numerical or categorical variables, accordingly.

Patients that met the inclusion and exclusion criteria will be asked to sign an informed consent followed by history-taking and blood sampling. The blood samples were then ordered for a routine hematology examination carried out using a hematology analyzer in the clinical pathology department. The measurement of CIMT will be carried by a cardiologist in the cardiovascular department using B mode ultrasound. The cardiologist will measure both of the carotid artery, and higher measurement of CIMT will be recorded.

The data were first exported to Microsoft Excel and then imported into Statistical Package for the Social Sciences (version 22) for quantitative statistical analysis software. All variables were subjected to descriptive statistics in order to describe the subject's frequency, percentage, means, and standard deviations prior to analysis. Homogeneity analysis was also performed in order to identify the factor of the confounding variable in the final analysis. Separate logistic regression models were performed to analyze the relationship between the main predictors and the main outcome. A separate analysis was conducted for each predictor. This study was approved by Health Research Ethics Committee in Moewardi General Hospital with the number: 1.320/XII/HREC/2020.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of CKD stage V
* on HD or CAPD based RRTs

Exclusion Criteria:

* cardiovascular, neoplastic, chronic inflammatory, or infectious disease
* usage of immunosuppressants or antiplatelet drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with a diagnosis of CKD stage V on HD or CAPD based RRTs from the department of renal-hypertension and hemodialysis unit in Moewardi General Hospital in Surakarta, Indonesia from January to July 2022.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Neutrophil-lymphocyte ratio (NLR) | Only in admission
  The absolute values of neutrophils that divided by the absolute values of lymphocytes
Platelet-lymphocyte ratio (PLR) | Only in admission
  The absolute values of platelet that divided by the absolute values of lymphocytes

CONTACTS AND LOCATIONS:
Locations (1):
- RS UNS (Universitas Sebelas Maret Hospital), Surakarta, Central Java, Indonesia